CLINICAL TRIAL: NCT00076947
Title: Evaluation of Tolerability and Safety of a Recombinant Purified HIV Envelope Vaccine
Brief Title: Safety of the EnvPro HIV Vaccine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P01AI045142-04 (NIH); EnvPro
Record Dates: First submitted 2004-02-06; First posted 2004-02-09 (Estimated); Last update posted 2008-03-21 (Estimated); Status verified 2005-03

CONDITIONS: HIV Infections
Keywords: HIV Preventive Vaccine; HIV Seronegativity; Protein
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: EnvPro

SUMMARY:
The purpose of this study is to determine the safety of a new HIV vaccine. The vaccine in this study is mixed with a chemical called alum to improve the body's response to the vaccine. Healthy adults who are not infected with HIV may participate in the study.

DETAILED DESCRIPTION:
EnvPro is a recombinant, purified envelope protein vaccine with an aluminum hydroxide (alum) adjuvant. Aluminum hydroxide is licensed as an adjuvant in other vaccines, such as the hepatitis B vaccine. This study will examine the safety and tolerability of EnvPro with alum adjuvant in healthy, HIV uninfected adults.

All participants in this study will receive vaccine injections in the upper arm muscle. Participants will receive a second vaccine injection eight weeks after the first injection. Blood tests will be performed at study visits before the vaccine is given, during the eight weeks between injections, and at selected times for up to three years after the vaccine is given.

ELIGIBILITY:
Inclusion Criteria:

* HIV uninfected
* Normal medical history and physical exam
* Normal complete blood count
* Normal liver function
* Normal renal function
* Normal serum creatine phosphokinase (CPK)
* Availability for at least 1 year follow-up

Exclusion Criteria:

* History of immunosuppressive illness, chronic illness, or use of any immunosuppressive medications
* Medical or psychiatric condition or occupational responsibilities which preclude compliance with the study
* Live attenuated vaccines within 60 days of study entry
* Use of experimental agents within 30 days of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2003-08

CONTACTS AND LOCATIONS:
Overall Officials: Karen Slobod, MD, Principal Investigator
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Background] Slobod KS, Lockey TD, Howlett N, Srinivas RV, Rencher SD, Freiden PJ, Doherty PC, Hurwitz JL. Subcutaneous administration of a recombinant vaccinia virus vaccine expressing multiple envelopes of HIV-1. Eur J Clin Microbiol Infect Dis. 2004 Feb;23(2):106-10. doi: 10.1007/s10096-003-1075-3. Epub 2004 Jan 20. PMID 14735404
- [Background] Brown SA, Stambas J, Zhan X, Slobod KS, Coleclough C, Zirkel A, Surman S, White SW, Doherty PC, Hurwitz JL. Clustering of Th cell epitopes on exposed regions of HIV envelope despite defects in antibody activity. J Immunol. 2003 Oct 15;171(8):4140-8. doi: 10.4049/jimmunol.171.8.4140. PMID 14530336
- [Background] Zhan X, Slobod KS, Surman S, Brown SA, Lockey TD, Coleclough C, Doherty PC, Hurwitz JL. Limited breadth of a T-helper cell response to a human immunodeficiency virus envelope protein. J Virol. 2003 Apr;77(7):4231-6. doi: 10.1128/jvi.77.7.4231-4236.2003. PMID 12634380
- See also: Click here for more information about the EnvPro study. — http://www.stjude.org/stjude/v/index.jsp?vgnextoid=f8e9588865e70110VgnVCM1000001e0215acRCRD&vgnextChannel=e5c0bfe82e118010VgnVCM1000000e2015acRCRD